CLINICAL TRIAL: NCT06627179
Title: A Two-Year Double-masked, Randomized, Sham-Controlled Study to Evaluate the Efficacy, Safety and Tolerability of Ultevursen in Subjects With Retinitis Pigmentosa (RP) Due to Mutations in Exon 13 of the USH2A Gene
Brief Title: Study to Evaluate Ultevursen in Subjects With Retinitis Pigmentosa (RP) Due to Mutations in Exon 13 of the USH2A Gene
Acronym: LUNA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratoires Thea (Industry)
Collaborators: Sepul Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SB-421a-006; 2024-515199-10-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-25; First posted 2024-10-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-07

CONDITIONS: Retinitis Pigmentosa (RP); Usher Syndrome Type 2; Deaf Blind; Retinal Disease; Eye Diseases, Hereditary; Eye Disorders Congenital; Vision Disorders
Keywords: Retinitis Pigmentosa; Usher Syndrome Type 2; Deaf Blind; USH2A; RP; Exon 13; RNA therapies; antisense oligonucleotide; exon skipping; LUNA; IVT; NSRP
MeSH Terms: conditions — Retinitis Pigmentosa; Usher Syndromes; Retinal Diseases; Eye Diseases, Hereditary; Eye Abnormalities; Vision Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ultevursen 180/60 μg (Experimental): Subjects will receive an intravitreal injection (IVT) of ultevursen with concentrations of 3.6 mg/mL for initial dose and 1.2 mg/mL for maintenance doses every 6 months thereafter through Month 18 (up to 4 doses).
  Interventions: Drug: Intravitreal Injection of Ultevursen
- Sham Procedure (Sham Comparator): Sham-procedure (no experimental drug administered)
  Interventions: Other: No intervention, will not receive any active study intervention

INTERVENTIONS:
Drug: Intravitreal Injection of Ultevursen — Up to 4 doses over a 24-month period
  Arms: Ultevursen 180/60 μg
Other: No intervention, will not receive any active study intervention — Sham-procedure (no experimental drug administered)
  Arms: Sham Procedure

SUMMARY:
The purpose of this Phase 2b study is to evaluate the safety and tolerability of ultevursen administered via intravitreal injection (IVT) in subjects with Retinitis Pigmentosa (RP) due to mutations in exon 13 of the USH2A gene. This is a multicenter Double-masked, Randomized, Sham-controlled study which will enroll 81 subjects.

DETAILED DESCRIPTION:
A total of eighty-one (81) RP subjects will be enrolled in this study, randomized in a 2:1 ratio to either ultevursen or sham procedure, respectively. Subjects randomized to the active treatment group will receive therapy with ultevursen administered via intravitreal (IVT) injection to the treatment eye (TE) on Day 1 and at Months 6, 12, and 18. Subjects randomized to sham will undergo a sham procedure in the TE at the corresponding timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. An adult (≥18 years) willing and able to provide informed consent for participation prior to performing any study related procedures
2. OR A minor (8 to <18 years) able to provide age-appropriate assent for study participation with a parent or legal guardian willing and able to provide written permission for the subject's participation prior to performing any study related procedures. An adult willing to comply with the protocol, follow study instructions, attend study visits as required and willing and able to complete all study assessments, in the opinion of the Investigator.

   OR A minor able to complete all study assessments and comply with the protocol and has a parent or caregiver willing and able to follow study instructions and attend study visits with the subject as required, in the opinion of the Investigator.
3. Both eyes exhibit clinical presentation consistent with RP involving Usher syndrome type 2 or NSRP based on ophthalmic, audiologic, or vestibular examinations. At screening, the Investigator will make the clinical diagnosis of "Usher syndrome type 2a," defined as RP with congenital hearing loss, or "non-syndromic RP," defined as RP without congenital hearing loss.
4. A molecular diagnosis of biallelic disease causing variants (pathogenic or likely pathogenic) in the USH2A gene where at least one of the variants is located on exon 13. A historic genotyping report from a certified laboratory is acceptable with Sponsor approval.
5. Clearly visible and measurable SD-OCT horizontal EZ width of ≥2.2 mm in both eyes based on the assessment of the CRC.
6. BCVA ≥55 letters based on ETDRS (equivalent to 20/80 based on Snellen notation, or logarithm of the minimum angle of resolution [logMAR] +0.6) in both eyes.
7. Impairment of VF as assessed by SP with a mean sensitivity greater than 4 decibels (dB) and less than 25 dB measured by a V target size in the TE at screening.
8. Mean sensitivity greater than 2 dB as determined by MP in the TE at screening.
9. Symmetry of baseline disease in both eyes, defined as the mean BCVA (based on ETDRS) of one eye within ≤10 letters of the mean BCVA of the other eye at screening.

Exclusion Criteria:

1. Presence of additional non-exon 13 USH2A pathogenic or likely pathogenic variant on the USH2A allele carrying the exon 13 mutation in subjects who have one exon 13 disease causing variant and one non-exon 13 disease causing variant.
2. Presence of additional non-exon 13 USH2A pathogenic mutation(s) on both USH2A alleles in subjects who have biallelic exon 13 mutations.
3. Presence of pathogenic or likely pathogenic variants in genes (other than the USH2A gene) which are known to be associated with other inherited retinal degenerative diseases or syndromes. Specifically, the presence of homozygous or compound heterozygous known disease-causing mutations in other genes involved in recessive retinal dystrophies, or the confirmed presence of a known single disease-causing variant in genes involved in dominant, X-linked, or mitochondrial retinal dystrophy genes is exclusionary.
4. At screening, the EZ horizontal or vertical width are outside the field of the SD-OCT scan based on the assessment of the CRC.
5. Presence of any significant ocular or non-ocular disease/disorder (including medication and laboratory test abnormalities) which, in the opinion of the Investigator may either put the subject at risk because of participation in the study, may impact the subject's ability to participate in the study, or may interfere with assessment of efficacy and safety in the study.
6. Presence of unstable concurrent cystoid macular edema (CME), or subject started on (or changed dose of) any medication for CME in the 3 months prior to enrollment. CME is allowed if stable for 3 months (with or without treatment). However, stable CME that disrupts the EZ width measurement, as determined by CRC, is an exclusion.
7. Any intraocular surgery within 3 months of study entry or any planned intraocular or peri-ocular surgery during the study. Subjects may be eligible after 3 months post-surgery as long as they have fully recovered, in the opinion of the Investigator.
8. Receipt of any IVT injection prior to study entry.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate efficacy after 24 months of treatment | 24 Months
  Annualized percent change from baseline in ellipsoid zone (EZ) width as measured by spectral-domain optical coherence tomography (SD-OCT) up to Month 24.

SECONDARY OUTCOMES:
Annualized change from baseline in static perimetry (SP) mean sensitivity | Month 24
Annualized change from baseline in microperimetry (MP) mean sensitivity | Month 24
Change from baseline in low luminance visual acuity (LLVA) using the Early Treatment Diabetic Retinopathy Study (ETDRS) chart | Month 24
Change from baseline in best-corrected visual acuity (BCVA) using the ETDRS chart | Month 24
Percent change from baseline in EZ area by SD-OCT | Month 24
Percent change from baseline in EZ width by SD-OCT | Month 24
Change from baseline in the Michigan Retinal Degeneration Questionnaire (MRDQ) for subjects ≥13 years of age | Month 24
  Michigan Retinal Degeneration Questionnaire (MRDQ) scores in central vision, color vision, contrast sensitivity, scotopic function, photopic peripheral vision, mesopic peripheral vision, and photosensitivity Unabbreviated scale title: Michigan Retinal Degeneration Questionnaire Minimum and Maximum values: -3 and +3 Higher scores indicate a worse outcome.
Change from baseline in the Michigan Vision-Related Anxiety Questionnaire (MVAQ) for subjects ≥13 years of age | Month 24
  Michigan Vision-Related Anxiety Questionnaire (MVAQ) scores in rod-function anxiety and cone-function anxiety.
  Unabbreviated scale title: Michigan Vision-Related Anxiety Questionnaire Minimum and Maximum values: -3 and +3 Higher scores indicate a worse outcome.
Frequency and severity of ocular and non-ocular adverse events (AEs) | Up to month 24
Systemic Exposure | Up to month 24
  Systemic serum concentration of ultevursen

CONTACTS AND LOCATIONS:
Locations (26):
- United States (10):
  - The University of California, San Francisco, San Francisco, California
  - Bascom Palmer Eye Institute/University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Massachusetts Eye and Ear, Boston, Massachusetts
  - University of Michigan- Kellogg Eye Center, Ann Arbor, Michigan
  - Casey Eye Institute, Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Scheie Eye Institute, Philadelphia, Pennsylvania
  - Retina Foundation of the Southwest, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Wisconsin- Madison, Madison, Wisconsin
- Ghent University Hospital, Ghent, Belgium
- Federal University of São Paulo - Hospital São Paulo (UNIFESP-HSP), São Paulo, Brazil
- Canada (2):
  - Hospital for Sick Children, Toronto, Ontario
  - McGill University Health Centre for Innovative Medicine, Montreal, Quebec
- Rigshospitalet and University of Copenhagen, Glostrup Municipality, Denmark
- France (2):
  - Hôpital Gui de Chauliac - CHRU de Montpellier - Maladies Sensorielles Génétique, Montpellier
  - Centre de maladies rares CHNO des Quinze Vingt, Paris
- Universitätsklinikum Tübingen, Tübingen, Germany
- Italy (2):
  - ASST Santi Paolo e Carlo Hospital, University of Milan, Milan
  - AOU Università degli Studi della Campania Luigi Vanvitelli, Napoli
- Netherlands (3):
  - Amsterdam University Medical Center - Locatie AMC, Amsterdam
  - Radboud Universitair Medisch Centrum, Nijmegen
  - Het Oogziekenhuis Rotterdam, Rotterdam
- United Kingdom (3):
  - Oxford Eye Hospital, Headington, Oxford
  - University of Edinburgh / NHS Lothian, Edinburgh
  - Moorfields Eye Hosptial, London

IPD SHARING:
Plan to Share IPD: No